CLINICAL TRIAL: NCT03254407
Title: Comparison of Cost-effectiveness Between Electronic Notes Versus Telephone Calls to Alert the Prescriber of a Possible IV to Oral Switch.
Brief Title: Switch Timely to Oral Medication
Acronym: STORM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, Thomas De Rijdt, Assistant-head of Pharmacy, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: S58200
Record Dates: First submitted 2017-05-01; First posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: IV Oral Switch; Appropriateness Review
Keywords: bioequivalent; IV/PO switch; appropriateness; clinical pharmacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening medical record (Other): Screening medical record for possible IV-PO switch Possbile IV/PO switch communicated to prescriber by phone or e-note
  Interventions: Other: Screening medical record

INTERVENTIONS:
Other: Screening medical record — Communicating possible IV/PO switch to prescriber by phone or e-note in medical record

SUMMARY:
The goal of this study compare the effectiveness of an electronic note versus a telephone call to alert the prescriber of a possible IV to oral switch. Secondary endpoints are the time-to-switch and the economic impact of earlier IV to oral switch.

DETAILED DESCRIPTION:
Methods

o Study design

A prospective, mono-centric, interrupted time series interventional study will be carried out starting in August 2015. Patients will be recruited hospital wide, except for patients admitted at the ICU or pediatric wards. The study protocol will be send for approval to the Clinical Trial Centre and Ethics Committee. Based on the NIH, Code of Federal Regulations Chapter 45-46, an exemption on informed consent is requested at Ethics Committee in order to prevent bias by informing physicians and/or patients; as there's only a suggestion to alter therapy to the treating physician and no clinical intervention is planned and data are processed anonymously and retrospectively, patient safety and patient rights are guaranteed. The study protocol will be registered in the public registry ClinicalTrials.gov.

o Inclusion and exclusion criteria and general assessment process

All prescriptions for levofloxacin (J01MA12), moxifloxacin (J01MA14), clarithromycin (J01FA09), fluconazole (J02AC01), clindamycin (J01FF01), acetaminophen (N02BE01), rifampicin (J04AB02), ornidazole (J01XD03) and metronidazole (J01XD01) in the hospitals CPOE from 01-08-2015 until 30-11-2015 for all hospitalized patients will be included.

The following prescription-related information will be requested from the HIS: unique hospitalisation number, patient name (needed for contact with prescriber), date of prescription, identification of prescriber, ward number, discipline, medication, route of administration, dose.

The sample size of the dataset is not limited in order to provide the maximum power to the study. The number of patients is estimated at 4000 per month.

o Building the dataset

A daily stored query, as presented in Figure 1, will the CPOE for therapies with at least one of the nine bio-equivalent drugs and fulfillment of the other criteria, such as presence of an order of a meal or prescription for other oral solid drugs and absence of a prescription of parenteral nutrition or an order for enteral feeding . The working procedure and the stored query are validated by 3 senior staff hospital pharmacists with expertise in the domain and approved by the Pharmacy&Therapeutics Committee (MFC).

The time scheme of the study is presented in Figure 2, and consists of the following blocks:

* Baseline monitoring periods: During month 1 and 3, the query will be run without intervention. The results of the query are captured in a database in order to have baseline data before starting both the intervention periods.
* Intervention period 1: During month 2, a team of trained staff pharmacists, who are assisted under close supervision by master students of the Faculty of Pharmaceutical Sciences, contact the prescribers by telephone, guided by the suggestions and information of the operating procedure. The number of contacted prescribers and their responses (acceptance or not) are recorded in the database. To do so, a standard operating procedure for telephone contact with the prescribers will be available for the co-investigators.
* Intervention period 2: During month 4, a computer algorithm will leave an electronic follow-up note suggesting the potential IV to oral switch, along with the argument to do so, in the medical record.

Due to dispensing of the medication and his interdisciplinary task in optimizing therapy the hospital pharmacist is related to the patient and has access to the necessary data; the pharmaceutical record is part of the patients' medical record. Nevertheless the access to the medical records is, as always, subject to approval by the medical council. Use of data is subject to a confidentiality agreement, an official confidentiality agreement between hospital and each co-investigator will be signed.

The solely intend of the access to the medical record is to gather data on the potential IV/PO switch and possible contra-indications. There will be no intervention in any way in the therapy nor the patient - physicians relationship. Reporting will be anonymous, never on an individual patient or physician.

Impact of initiation time of the study At the University Hospitals Leuven, August is the moment where most new prescribers enter the hospital. To avoid bias from this prescriber switch, the switch period is excluded from the timing. Therefore, in concrete, baseline monitoring period 1 will be started up in September 2015.

Avoidance of potential bias To avoid learning bias from the prescribers, a wash-out period is included before each intervention period. A poster on possible IV-PO switch will distributed in the hospital and published on the intranet webpage at the start of each period of the study.

o Analysis of database

General analysis of the database will be done in Microsoft Access 2013. More in detail, descriptive statistics will be carried out using appropriate parametric or non- parametric tests (Student t-test, Mann-Whitney U-test or Chi square, based on distribution of data) to describe the demographics of the included patients.

Statistical analysis will be carried out in SPSS or SAS by the investigator in collaboration with L-Biostat (KU Leuven).

o Pharmacoeconomic analysis

Based on the dataset (time-to-switch and price of medication) the potential cost-saving from a healthcare payer perspective will be calculated using the list price at 01-11-2015 of the involved medication. Cost-avoidance due to lesser infections or lesser length of stay cannot be calculated with this dataset.

ELIGIBILITY:
Inclusion Criteria:

* Therapy with prescriptions for levofloxacin (J01MA12), moxifloxacin (J01MA14), clarithromycin (J01FA09), fluconazole (J02AC01), clindamycin (J01FF01), acetaminophen (N02BE01), rifampicin (J04AB02), ornidazole (J01XD03) and metronidazole (J01XD01) in the hospitals CPOE from 01-08-2015 until 30-11-2015 for hospitalized patients.

Exclusion Criteria:

* Therapy prescribed in PDMS (in casu: ICU)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8000 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the type of alert | 4 months - August till November 2015 - calculated after each from 4 periods (=months)
  Difference in number of switches and time to swich between electronic note and telephone alert of the prescriber.

SECONDARY OUTCOMES:
The number of possible IV/PO switches, per discipline and per type of product | 4 months - August till November 2015 - calculated after each from 4 periods (=months)
  number of potential IV to oral switches
Pharmacoeconomic impact of the intervention on time to switch | 4 months - August till November 2015 - calculated after each from 4 periods (=months)
  Cost saving of switching to less expensive oral medication and cost saving due to lesser adverse events in relation to the cost of running the IV/oral switch service. Delta time to switch multiplied by days of inapproriate IV therapy --> savings in euro
Evidence and motivation for overruling the switch | 4 months - August till November 2015 - calculated after each from 4 periods (=months)
  Reasons and evidence background of the reasons for not following the advice to switch. descriptive.
Learning curve over time and this for both methods of alerting on possible IV/PO switches | 4 months - August till November 2015 - calculated after each from 4 periods (=months)
  Can there be a bias from a learning effect. Measured as time to switch in control and washout periods.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas De Rijdt, PharmD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No